CLINICAL TRIAL: NCT07347275
Title: A Multi-Centre, Randomised, Controlled Trial to Evaluate the Efficacy of DIALIVE 2.0, a Liver Dialysis Device, for the Treatment of Acute-on-Chronic Liver Failure (ACLF) A-TANGO Grade 2-4 Compared to Standard of Care (SoC)
Brief Title: A Novel Extracorporeal Liver Support Therapy In ALCF and to Evaluate the Efficacy of DIALIVE 2.0, a Liver Dialysis Device.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yaqrit Ltd (Industry)
Collaborators: University College, London (Other); King's College Hospital NHS Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YAQ002-ES-1; 206537 (Other Grant/Funding Number: NIHR); CI/2025/0075/GB (Other: MHRA); 353362 (Other: IRAS ID)
Record Dates: First submitted 2025-12-11; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute-on-Chronic Liver Failure (ACLF); Liver Cirrhosis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Cirrhosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Seventy-two evaluable participants will be randomised 1:1 to receive either Standard of care (SoC) or Standard of care (SoC) + DIALIVE 2.0. We will use stratified randomisation with 60% of participants presenting with A-TANGO Acute-on-Chronic Liver Failure (ACLF) grade 2 and 40% with grades 3 or 4 in each treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Standard of Care (Investigator Choice)
  Interventions: Other: Standard of Care (Investigator Choice)
- Treatment Group (Experimental): DIALIVE 2.0 liver dialysis Device plus available Standard of Care (Investigator Choice)
  Interventions: Other: Standard of Care (Investigator Choice); Device: DIALIVE 2.0 liver dialysis Device plus available Standard of Care

INTERVENTIONS:
Other: Standard of Care (Investigator Choice) — Standard of care as per Investigator discretion
Device: DIALIVE 2.0 liver dialysis Device plus available Standard of Care — DIALIVE 2.0 liver dialysis Device plus available Standard of Care
  Arms: Treatment Group

SUMMARY:
This study is intended to demonstrate the efficacy and safety of the DIALIVE Liver Dialysis Device when incorporated into the standard management plan for participants with A-TANGO ACLF grade 2-4.

A total of 72 evaluable participants, aged 18-70, will be enrolled in up to 12 clinical centres in the United Kingdom. Participants must have a history of liver cirrhosis and a deterioration within four weeks due to a precipitating event, leading to A-TANGO ACLF grade 2-4. Multicenter, individually randomised, controlled, open-label, parallel group trial using double-arm design. The control group will receive SoC for participants with ACLF. The DIALIVE 2.0 treatment group will receive SoC with the addition of up to 7 (seven) daily DIALIVE 2.0 treatment sessions within the 10-day treatment window. Seventy-two participants with ACLF (60% A-TANGO ACLF grade 2 at randomisation, and 40% A-TANGO ACLF grade 3 & 4 at randomisation) will be randomised 1:1 to receive either SoC or SoC + DIALIVE 2.0. This allows for 5% loss due to drop-out, and 5% censoring due to liver transplantation within 28 days. All randomised participants will be included in the intention to treat (ITT) analysis while all participants that receive at least one treatment cycle will be used for the safety population. For each participant, the study duration will be up to 105 days (screening: 5 days; treatment up to 10 days; follow up 90 days).

The total study duration is estimated to be approximately 18 months from screening of first participant until study completion of the last participant.

DETAILED DESCRIPTION:
DIALIVE 2.0 is an innovative liver dialysis device that specifically targets the underlying mechanisms of acute-on-chronic liver failure.

The novelty of DIALIVE 2.0 lies in the combined use of a commercially available high cutoff filter and an extracorporeal endotoxin adsorber integrated into a hemofiltration and plasmapheresis platform. This allows controlled extracorporeal circulation of the participant's blood, during which the system removes dysfunctional, toxin-bound albumin and circulating endotoxins, while simultaneously replenishing functional albumin. The result is a comprehensive therapeutic approach that addresses both immune dysregulation and impaired albumin detoxification capacity in acute-on-chronic liver failure. This treatment concept is referred to as Selective Plasma filtration, Endotoxin Adsorption, and Albumin Replacement (SPEAR), reflecting the three core processes that underpin DIALIVE 2.0's mode of action.

DIALIVE 2.0 is delivered as a daily treatment lasting six to eight hours, with a plasma filtration dose equivalent to 5% of the participant's ideal body weight. Albumin is replaced at a dose of one gram per kilogram of body weight using a 20% human albumin solution to offset albumin losses and maintain oncotic pressure. To address coagulation factor depletion observed in preclinical studies (see Investigators Brochure), one unit of fresh frozen plasma is administered at the end of each session to restore haemostatic balance.

The DIALIVE 2.0 system includes the following components:

* Medica FRACTIOsmart Small 1.0 haemodialyser with a high cut-off membrane (150 to 200 kilodaltons), used for the removal of albumin-bound toxins and medium-sized inflammatory molecules. This component is commercially available under European certification MDR 00048-A.
* Alteco® Medical LPS Adsorber, an extracorporeal filter designed for the selective removal of circulating endotoxin in conditions where endotoxemia is suspected or confirmed. This is a commercially available device certified under CE 0402, (awaiting MHRA registration).
* Medica AFERsmart Plus™ System, a plasmapheresis platform that controls flow rates, treatment duration, and pressure regulation. This is commercially available, and CE marked under number 0476.
* Medica AFERsmart Standard TPE Line, a sterile, CE-marked disposable tubing set compatible with the AFERsmart Plus device.
* Male to male tubing set, and absorber connector, (pending commercial approval).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years, with a diagnosis of ACLF grade 2-4 (according to A-TANGO ACLF criteria, APPENDIX 1)
* ACLF non-responsive to SoC for up to 48 hours prior to developing grade 2-4 ACLF.
* Inclusion within 10 days from the onset of A-TANGO ACLF grade ≥ 2.

Exclusion Criteria:

* A-TANGO ACLF grade ≥2 for more than 10 days prior to inclusion
* Pregnancy
* Co-infection with HIV and AIDS defining illness i.e. CD4+ T-cell count below 200 cells/µL, a CD4+ T-cell percentage of total lymphocytes of less than 15%, or one of the defining illnesses such as PCP, Kaposi's sarcoma, CMV, Candidiasis etc.
* Bacterial infection or sepsis unresponsive to treatment with antimicrobials for 48 hours indicated by (a) persistent pyrexia (b) rising white cell count, creactive protein and lactate (c) persistently positive cultures for bacteria or fungi and/or (d) worsening clinical state indicated by escalating requirement for fluid resuscitation, increasing vasopressors requirements or increasing organ support.
* Invasive fungal infection (clinical or radiological evidence, not solely biomarker positivity such as BDG or galactomannan)
* Acute or sub-acute liver failure in the absence of cirrhosis
* Post-hepatectomy liver failure or primary non-function following transplantation
* Previous liver transplant
* Severe thrombocytopaenia (absolute platelet count <20,000/mm3 at screening) or evidence of rapid decline in platelet count (> 50% reduction within the preceding 24 hrs)
* INR >3.0, unless sustained correction for >24 hours following FFP/PCC treatment
* Severe disseminated intravascular coagulopathy (DIC)
* Persistent haemodynamic instability as defined by:

  (i) Norepinephrine(NE) dose >0.5µg/kg/min, or, (ii) If a second pressor is used, a composite Norepinephrine equivalence index (NEEI) of dose >0.5µg/kg/min (iii) Arterial lactate level >4mmol/L despite 24 hours of adequate fluid resuscitation and pressor therapy
* Severe respiratory failure: PaO2/FiO2 (P/F) ≤ 200 mmHg or 27kPa
* Established on renal replacement therapy for longer than 24 hours prior to inclusion
* A-TANGO WCC ACLF score >64 (APPENDIX 1)
* Significant and/or uncontrolled bleeding (participants can be enrolled 48 hours after bleeding is controlled)
* Active or prior history of non hepatic malignancy unless adequately treated or in complete remission for five or more years
* HCC outside of Milan criteria.
* Acute, extensive, portal vein thrombosis extending to and occluding superior mesenteric vein
* Major systemic illness, aside from liver disease, that in the opinion of the investigator would preclude the participant from participating in the study (e.g. coronary artery disease, cerebrovascular disease, chronic pulmonary disease, chronic kidney disease, serious psychiatric disease)
* Pre-existing chronic kidney disease (CKD) defined as eGFR (estimated glomerular filtration rate) <30 mL/min for 3 months or longer prior to screening
* Severe frailty (Clinical Frailty Scale, CFS>5)
* Severe malnourishment (BMI<18)
* Participants not considered appropriate for full active treatment including organ support
* Participants who have a "do not attempt cardio-pulmonary resuscitation" order in place
* Any participant who has received an investigational drug or device within 30 days, or who is scheduled to receive another investigational drug or device during the course of the study (concomitant observational studies are allowed)
* Uncontrolled seizures
* Evidence of new intracranial pathology such as cerebral hemorrhage or infarction.
* Participants diagnosed with Creutzfeldt-Jakob disease.
* Participants unable to consent for themselves, unless a legal representative/consultee is appointed and approved as dictated by local and national legislation.
* Known allergy to heparin, or type II thrombocytopaenia caused by heparin (HIT syndrome type II).
* In the opinion of the investigator, recruitment to the the study would be unsafe for the participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Resolving ACLF symptoms using DIALIVE 2.0 treatment | From Baseline to within 10 Days
  DIALIVE 2.0 treatment plus SoC is safe and provides a significant increase in the proportion of participants resolving ACLF within 10 days of treatment.

SECONDARY OUTCOMES:
Comparison of DIALIVE 2.0 treatment along with Standard of Care (SoC) & patients treated with only SoC. | Post Enrollment to 28 and 90 days
  Increase in transplant-free survival post enrolment
DIALIVE 2.0 plus standard of care (SoC) does not increase the incidence of SAEs | From baseline to Day 28 & Day 90
  Decrease incidences of related SAEs
Comparison of DIALIVE 2.0 treatment along with Standard of Care (SoC) & patients treated with only SoC. | baseline to day 28.
  Increase in predicted six-month and one-year survival rate of the patients.
Comparison of DIALIVE 2.0 treatment along with Standard of Care (SoC) & patients treated with only SoC. | Day 0 to 28 days
  decrease time to discharge from ICU and/or hospital.
Comparison of DIALIVE 2.0 treatment along with Standard of Care (SoC) & patients treated with only SoC | Baseline to Day 28
  Increase the proportion of participants that have resolved individual organ failures
Comparison of DIALIVE 2.0 treatment along with Standard of Care (SoC) & patients treated with only SoC. | Baseline to Day 10
  resolution of A-TANGO ACLF grade 2-4 to absence of ACLF